CLINICAL TRIAL: NCT00590915
Title: Erwinase Master Treatment Protocol
Acronym: EMTP
Status: No longer available | Type: Expanded Access
Sponsor: Phoenix Children's Hospital (Other)
Collaborators: Fisher Bioservices (Industry); Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: Erwinase; IND-290; NCT01009164 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2012-04

CONDITIONS: Leukemia, Acute Lymphoblastic; Acute Lymphoid Leukemia
Keywords: ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — asparaginase erwinia chrysanthemi recombinant; Asparaginase

INTERVENTIONS:
Drug: Erwinia L-asparaginase — Substitute Erwinia L-asparaginase 25,000 international units per meters squared, IM every other day (including weekends and holidays) x 6 doses for each dose of PEG-asparaginase that is replaced.
  NOTE: Erwinia L-asparaginase dosing to replace native E.coli L-asparaginase varies; consult protocol for specifics.
  Other Names: Erwinase

SUMMARY:
The purpose of this study is to make Erwinase available to patients with acute lymphoblastic leukemia (ALL) who have had previous allergic reactions to certain formulations of L-asparaginase.

ELIGIBILITY:
Inclusion Criteria:

* Patient must give written informed consent to receive Erwinase.
* Patient must be treated for acute lymphoblastic leukemia.
* Patient must have either systemic hypersensitivity reactions to native (Elspar) or pegylated E.coli asparaginase (Oncaspar). This includes patients with generalized rash with or without anaphylactic symptoms, or patients with previously documented local or systemic reactions to E.coli derived L-asparaginase.

Exclusion Criteria:

* Previous allergic reaction to Erwinia L-asparaginase (Erwinase)
* Previous acute pancreatitis
* Pregnant or lactating woman

Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- See also: Phoenix Children's Hospital — http://www.phoenixchildrens.com
- See also: EUSA Pharma (US), Inc.- manufacturer of Erwinase — http://www.eusapharma.com